CLINICAL TRIAL: NCT04922294
Title: Cardiometabolic Disease Staging System to Improve Medical Management of Obesity and Diabetes in Primary Care Settings
Brief Title: Implementation of a Cardiometabolic Disease Staging System in Primary Care
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tapan Shirish Mehta, Associate Professor, Director of Research, University of Alabama at Birmingham
Other Study IDs: IRB-300003559
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Diabetes; Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Overweight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical decision support system — To develop a clinical decision support system based on a published cardiometabolic disease staging system.

SUMMARY:
The aim of this study is to develop a clinical decision support system (CDSS) that incorporates obesity management guidelines and treatment options for use by physicians and, potentially, patients based on a cardiometabolic disease staging system. This CDSS will be designed using primary care provider input through a qualitative approach to explore physician preferences for the appearance, electronic location, treatment options, referrals, accessibility and other user requirements of the CDSS.

DETAILED DESCRIPTION:
To provide appropriate medical management of obesity and facilitate the diabetes risk assessments of people with excess adiposity, a comprehensive staging system that establishes five stages of cardiometabolic disease risk-the cardiometabolic disease staging system (CMDS) has been developed. This staging is based on Adult Treatment Panel III metabolic syndrome risk factors to guide decision making for selection of treatment modality and intensity in the management of obesity. Hence, the study hypothesis is that providing CMDS to PCPs through a CDSS for medical management of obesity can aid in reducing the barriers of obesity and diabetes treatment at the PCP-level and improve the quality of obesity and diabetes care. In this pilot and feasibility study, investigators will implement an early-phase CDSS in a pragmatic PCP setting to assess the uptake and acceptability of CDSS delivered to PCPs implementing CMDS at the point of care, and collect pilot data to assess change in patient engagement and satisfaction.

Investigators will conduct initial focus groups with PCPs and a series of iterative design steps targeting PCP and patient needs. These qualitative interviews would be used to determine the initial set of requirements and prototypes of the user interfaces and notifications.

ELIGIBILITY:
Inclusion Criteria:

* Primary care physicians employed at the University of Alabama at Birmingham

Exclusion Criteria:

* Physicians ≥19

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care physicians employed at the University of Alabama at Birmingham within the Primary Care or Family Medicine departments
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Implementation preferences | Over one hour interviews or focus groups
  Preferences for implementation and development of a cardiometabolic disease staging system for a clinical decision support system as identified by clinicians during qualitative focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Tapan S Mehta, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No